CLINICAL TRIAL: NCT06800209
Title: Pain Reprocessing Therapy in Post-Operative Knee Pain
Acronym: REJOICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Hospital for Special Surgery, New York (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-2140; 24-2140 (Other: COMIRB)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pain, Chronic; Knee Pain Chronic
Keywords: chronic pain; Pain Reprocessing Therapy; knee pain; total knee replacement; Total Knee Arthroplasty; mind-body; mindfulness; TKA; PRT
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment will be completed via automated transmission of a REDCap link, and as such is inherently blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain reprocessing therapy (PRT) (Experimental): PRT has five components: 1) education about the origin of pain in the brain, its reversibility, and the pain-fear cycle; 2) reinforcing education using personal biography; 3) "somatic tracking" of pain through mindfulness and reappraisal of pain sensations as non-dangerous; 4) lowering the level of personal threat that may trigger pain sensation; and 5) inducing positive affect in periods of pain. Patients will attend eight 50-minute, therapist-led sessions. Pacing will be weekly, for approximately eight weeks.Treatment will be provided by experienced PRT clinicians. All PRT sessions will be remotely delivered.
  Interventions: Behavioral: Pain reprocessing therapy (PRT)
- Usual Care (Other): Participants will be asked to continue whatever they are already doing to care for their knee pain. Length of the usual care condition will be eight weeks, the expected completion time of the PRT arm.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Pain reprocessing therapy (PRT) — A promising new psychotherapy for chronic pain.
  Arms: Pain reprocessing therapy (PRT)
Other: Usual care — Participants will be asked to continue to do whatever they are currently doing to manage their pain.
  Other Names: Treatment as usual
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to learn whether Pain Reprocessing Therapy (PRT) can help adults with knee pain after knee replacement surgery. The study is comparing PRT to usual care (the regular treatment people get after surgery) to see which works better for relieving pain.

The main questions the study aims to answer are:

1. Does PRT help lower pain in people who have chronic knee pain after knee surgery?
2. How do the effects of PRT compare with usual care in terms of pain relief and other factors such as anxiety, depression, and sleep?
3. How does PRT impact the brain?

Participants will:

1. Be randomly assigned to receive either PRT or usual care.
2. Complete questionnaires about their pain and health.
3. If in the PRT group, have eight weekly therapy sessions over video calls with a therapist.
4. If interested, may also take part in an optional EEG test to measure brain activity related to pain.

DETAILED DESCRIPTION:
Investigators recently developed a novel psychological treatment called Pain Reprocessing Therapy (PRT). Using a combination of cognitive, exposure-based, and somatic psychotherapy techniques, PRT aims to promote patients' reconceptualization of pain as due to reversible, non-dangerous brain activity rather than peripheral pathology. Critically, PRT aims to reduce or eliminate pain, rather than merely increase functioning.

In the first trial of PRT (N = 151), 66% of patients randomized to PRT were pain-free or nearly pain-free at post-treatment, compared to fewer than 20% of those in the placebo and usual care control groups. This trial was limited to chronic back pain and the efficacy and mechanisms of PRT for chronic post-operative knee pain are unknown. Additionally, how the effects of PRT will generalize to telehealth treatment is not known.

Developing scalable, effective, non-pharmacological chronic pain treatments and testing their efficacy in underserved populations is an urgent societal need. Accordingly, this study also tests a remotely delivered PRT intervention.

Aim 1 of this study is to test the comparative efficacy of PRT vs. usual care on pain intensity and other pain-related outcomes at post-treatment and longitudinal follow-up.

Aim 2 of this study is to test hypothesized psychological and neurobiological mechanisms of PRT with mediation analyses and longitudinal EEG neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients are deemed eligible at 3 months post-operatively if: The patient completed a primary knee replacement [surgery completed without complication and patient exhibits full mechanical joint function, as determined by the treating physician (good range of motion, stability, and wound healing; absence of swelling)] and patient reports last week average knee pain ≥ 4 of 20 and at least two questions rated 'moderate' on A 12-item shortened version (ShortMAC) of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
* Reported pre-operative chronic knee pain of at least 6 months duration prior to surgery
* The procedure was a primary (not a revision) knee replacement
* Proficient in English

Exclusion Criteria:

* Patients who are not willing to participate in a telehealth visit.
* Patients with pre-op chronic pain but who do not have post-operative pain after the three month time period.
* Active suicidal ideation with intent, recent history of suicide attempt, or self-harm behaviors within the past 5 years (including non-suicidal self-harm).
* Recent history of inpatient psychiatric hospitalization within the past 5 years.
* Active, current psychosis or mania.
* Active, current substance abuse, or problems with substance abuse within the past 2 years.
* Instability in living conditions or major interfering life events:

  * Major surgery or other major medical event planned in coming 6 months.
  * Uncertain whether they will have suitable conditions for telehealth appointments over the next 2 months, including access to a computer or tablet, reliable high-speed internet, and a quiet, comfortable room that is consistently available.
  * Major, interfering changes in employment or housing anticipated over the next 6 months.
* Neurological conditions (e.g., Alzheimer's, dementia, mild cognitive impairment, Huntington's disease, multiple sclerosis, cerebral palsy). This will be case-by-case decision made by PI to determine if the condition may interfere with treatment and warrant exclusion.
* Self-reported diagnosis of an autoimmune disease (e.g., rheumatoid arthritis, polymyalgia rheumatica, scleroderma, lupus, polymyositis, or another autoimmune disorder).
* Currently or plan to be involved in lawsuits related to pain in next 6 months, currently or plan to apply for any disability payments related to the pain in next 6 months, or received legal settlement or other disability payments related to the pain over past 2 years.

EEG Exclusion Criteria (patients can still be enrolled as long as they meet all other eligibility criteria; however, they will not undergo EEG testing):

* Are unable or uncomfortable with completing a dry cap EEG.
* Has had a history of abnormal EEGs.
* Had bilateral TKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Approximately 12, 18, and 26 weeks post-randomization
  Last-week average pain intensity is assessed using the 5-item pain subscale of the 12-item shortened version (ShortMAC) of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The ShortMAC assesses pain severity and its impact on functioning. It consists of 12 total items, including 5 pain items and 7 pain interference items. The 5 pain items measure pain on a scale of 0-4, with 0 indicating no pain and 4 indicating extreme pain.

SECONDARY OUTCOMES:
Pain interference | Approximately 12, 18, and 26 weeks post-randomization
  Pain interference is assessed using the 7-item pain interference subscale of the 12-item shortened version (ShortMAC) of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The ShortMAC assesses pain severity and its impact on functioning. It consists of 12 total items including 5 pain items and 7 pain interference items. The 7 pain interference items measure pain interference in the last week on a scale of 0-4, with 0 indicating no difficulty and 4 indicating extreme difficulty or inability to perform an activity.
Depression | Approximately 12, 18, and 26 weeks post-randomization
  Depression is assessed using the 8-item depression subscale of the Patient-Reported Outcome Measurement Information System Short Form (PROMIS-SF). The PROMIS scale as a whole monitors the physical, mental, and social health of adults and children. Each item in the PROMIS-SF depression subscale is rated on a 5-point scale of 1 (never) to 5 (always).
Anxiety | Approximately 12, 18, and 26 weeks post-randomization
  Anxiety is assessed using the 8-item anxiety subscale of the Patient-Reported Outcome Measurement Information System Short Form (PROMIS-SF). The PROMIS scale as a whole monitors the physical, mental, and social health of adults and children. Each item in the PROMIS-SF anxiety subscale is rated on a 5-point scale of 1 (never) to 5 (always).
Fatigue | Approximately 12, 18, and 26 weeks post-randomization
  Fatigue is assessed using the 8-item sleep disturbance subscale of the Patient-Reported Outcome Measurement Information System Short Form (PROMIS-SF). The PROMIS scale as a whole monitors the physical, mental, and social health of adults and children. 7 of the 8 items in the PROMIS-SF sleep disturbance subscale are rated on a 5-point scale of 1 (not at all) to 5 (very much) while 1 item is rated on a 5-point scale of 1 (very poor) to 5 (very good).
Opioid Use | Approximately 12, 18, and 26 weeks post-randomization
  Opioid Use is assessed via patient-reported medication logs

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified project data publicly under Data Use Agreements that safeguard individual participant confidentiality and privacy. The study will produce the following types of data. All data will be available for sharing, except where noted, upon the date of the online publication of the results of the primary study aims:
  * Patient-reported outcomes: All patient-reported outcomes will be de-identified and shared in raw form.
  * Measures of treatment engagement: De-identified values (e.g., number of treatment sessions attended) will be shared in raw form.
  * EEG patient-level summary statistics (de-identified).
Time Frame: Complete, clean, de-identified copies of the data components described above, along with data dictionaries and metadata, will be publicly posted along with data use agreements by the online publication date of the primary aims in a peer-reviewed journal.
Access Criteria: Data Use Agreements will ask users to not attempt to re-identify participants, either by merging in administrative, census, medical, or other data, or by using a software program that might re-identify participants.
  Investigators will consult, as needed, with Cornell Data Services (CDS), formerly known as Cornell Research Data Management Service Group (RDMSG). As described in the Cornell Roybal Center's overall data-sharing plan, through the Cornell Roybal Center Investigator Development Program, investigators will have access to instruction and assistance to address requests for information that ensure research transparency and reproducibility: documentation on study aims; hypotheses/research questions; variable sources (e.g., outcome variables, covariates); measure/index construction; and publication information.